CLINICAL TRIAL: NCT05971160
Title: Creating Access to Resources and Economic Support
Acronym: CARES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00113319; R01MD016755 (NIH)
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Psychological Distress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (Active Comparator): Monthly financial education videos and one-time microgrant
  Interventions: Behavioral: Financial education videos; Other: Microgrant
- Monthly microgrants (Active Comparator): Monthly financial education videos and monthly microgrants
  Interventions: Behavioral: Financial education videos; Other: Microgrant
- Monthly microgrants plus peer mentoring (Active Comparator): Monthly financial education videos, monthly microgrants, and peer mentoring support
  Interventions: Behavioral: Financial education videos; Other: Microgrant; Behavioral: Peer mentoring

INTERVENTIONS:
Behavioral: Financial education videos — Brief videos providing structured information on managing one's money
Other: Microgrant — $150 stipend
Behavioral: Peer mentoring — One-on-one structured mentoring sessions with a trained peer
  Arms: Monthly microgrants plus peer mentoring

SUMMARY:
The goal of this study is to test the ability of small grants and/or peer support to improve mental health among transgender people experiencing material hardship. The main questions the study will answer are:

1. Do microgrants with or without peer mentoring improve mental health?
2. Do microgrants with or without peer mentoring improve mental health by reducing material hardship and/or increasing a sense of community connection?

Researchers will compare mental health outcomes among three groups of participants:

A. Participants who receive one small grant and monthly financial education videos B. Participants who receive a small grant every month and monthly financial education videos for a total of 6 months.

C. Participants who receive a small grant every month, peer mentoring support, and monthly financial education videos for a total of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* gender identity different from sex assigned on original birth certificate
* access to a mobile phone or email
* score > 0 on the material hardship index

Exclusion Criteria:

* inability to provide informed consent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender different from sex assigned at birth
Enrollment: 360 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in psychological distress, as measured by Kessler 6 | Baseline, 6 months, 12 months
  Kessler 6 is a 6-item scale with each item scored from 0-4 for a total score range from 0-24, with higher scores indicating greater psychological distress.

SECONDARY OUTCOMES:
Change in substance use, as measured by the Drug Abuse Screening Test (DAST-10) | Baseline, 6 months, 12 months
  DAST-10 is a 10-item scale with with one one point for each "yes" response for a total score range from 0-10, with higher scores indicating more problematic substance use

CONTACTS AND LOCATIONS:
Overall Officials: Tonia C. Poteat, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University (online recruitment), Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share data via one of the NIH repositories listed by the Trans-NIH BioMedical Informatics Coordinating Committee (BMIC). The final available dataset from this proposed research will include self-reported demographic, psychosocial, and behavioral data from quantitative surveys. No personal identifiers will be included with the final available dataset.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available 12 months after publication of primary study findings.
Access Criteria: In accordance with the NIH Data Sharing Policy and Implementation Guidance, the investigators will make the data and supporting information available to users under a data-sharing agreement that provides for: (1) complete protection of human subjects training and a commitment to research ethics; (2) a commitment to using the data only for research purposes and not to identify an individual participant; (3) a commitment to securing the data using appropriate technology, and (4) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Derived] Poteat TC, Reisner SL, Wirtz AL, Mayo-Wilson LJ, Brown C, Kornbluh W, Humphrey A, Perrin N. A Microfinance Intervention With or Without Peer Support to Improve Mental Health Among Transgender and Nonbinary Adults (the Creating Access to Resources and Economic Support Study): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Aug 26;13:e63656. doi: 10.2196/63656. PMID 39186770

DOCUMENTS (1):
  • Informed Consent Form (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/60/NCT05971160/ICF_000.pdf